CLINICAL TRIAL: NCT00336895
Title: Conversion of CellCept to Myfortic: A Prospective Study on the Tolerability and Safety of Myfortic in Liver Transplant Recipients
Brief Title: Conversion of CellCept to Myfortic: A Prospective Study in Liver Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Roberto Lopez, MD, Assistant Professor of Surgery, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERL080A-US27
Record Dates: First submitted 2006-06-12; First posted 2006-06-14 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Immunosuppression
Keywords: Liver transplantation; mycophenolate mofetil; gastrointestinal; adverse effects
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liver Transplant Subjects (Experimental): All subjects in this study will receive Myfortic 360mg or 720 mg BID for 90 days.
  Interventions: Drug: Myfortic

INTERVENTIONS:
Drug: Myfortic — Myfortic 360mg or 720 mg BID for 90 days.

SUMMARY:
The objective of this study is to determine the tolerability and safety of Myfortic in liver transplant patients. Patients receiving CellCept who have GI side effects will have CellCept discontinued and changed to Myfortic (Myfortic is a new drug similar to CellCept, except it is enteric-coated). Our hypothesis is that Myfortic has less GI side effects and will, therefore, be tolerated better than CellCept and also that Myfortic will have a comparable effectiveness to CellCept.

DETAILED DESCRIPTION:
This is a prospective, single center, open-label, safety and tolerability study on the use of Myfortic after liver transplantation. Adult liver transplant patients who are experiencing GI symptoms (nausea, vomiting, diarrhea, abdominal discomfort/pain, dyspepsia) attributable to CellCept are eligible to enter the study. CellCept will be discontinued and replaced with Myfortic. The duration of the study will be 3 months, and during this time, we will assess the incidence and severity of GI adverse events, the incidence and severity of bone marrow suppression (leukopenia), and the incidence of cytomegalovirus (CMV) infection or disease in patients receiving Myfortic.

ELIGIBILITY:
Inclusion Criteria:

* ALL patients will be adult liver transplant recipients, males or females, 18-80 years of age
* Patients currently receiving tacrolimus or cyclosporine with or without corticosteroids as part of their immunosuppressive regimen
* Patients must be receiving CellCept and must have attributable G.I. symptoms (nausea, vomiting, diarrhea, abdominal discomfort/pain, dyspepsia)
* Patients must be more than 30 days post-transplant to be eligible
* Females of childbearing potential must have a negative serum pregnancy test prior to the inclusion period

Exclusion Criteria:

* Multi-organ transplant patients
* HIV positive patients.
* Living-related liver transplant recipients
* Pregnant patients
* Patients with a history of extra-hepatic malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin
* Patients with thrombocytopenia (<50,000/mm3), with an absolute neutrophil count of <1,000/mm3 and/or leukocytopenia (<2,000/mm3), and/or hemoglobin <7.0 g/dL prior to enrollment
* Patients with a G.I. clinical problem at the time of enrollment (e.g. CMV infection or disease, C. difficile colitis, active peptic ulcer disease, gastroenteritis, inflammatory bowel disease)
* Presence of clinically significant infection requiring continued therapy or uncontrolled diabetes mellitus
* Evidence of drug and/or alcohol abuse
* Decisionally impaired subjects who are not medically or mentally capable of providing consent themselves

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E de Vera, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 participants were screened only 29 participants were enrolled
Period: Overall Study
Arm/Group | Liver Transplant Subjects
Started | 30
Completed | 26
Not Completed | 4
Not completed — diarrhea | 1
Not completed — nausea and upset stomach | 1
Not completed — Physician Decision | 1
Not completed — screen failed | 1

BASELINE CHARACTERISTICS:
Population: 30 potential participants were screened but only 29 enrolled.
Arm/Group | Liver Transplant Subjects
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (13.0)
Gender [Count of Participants; unit: Participants]
  Female | 13
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 29
Abdominal Pain- screening [Mean (Standard Deviation); unit: units on a scale] — The gastrointestinal Symptom Rating Scale (GSRS) is a validated scale, the items range from 1= No discomfort at all to 7= Very severe discomfort.
  The scale ranges from a minimal value of 3 ( No discomfort at all) to a maximum of 21 ( Very severe discomfort)
  units on a scale | 10.7778 (5.09399)
Reflux screening [Mean (Standard Deviation); unit: units on a scale] — The gastrointestinal Symptom Rating Scale (GSRS) is a validated scale, the items range from 1= No discomfort at all to 7= Very severe discomfort.
  The scale ranges from a minimal value of 2 ( No discomfort at all) to a maximum of 14 ( Very severe discomfort)
  units on a scale | 5.0000 (3.67423)
Indigestion screening [Mean (Standard Deviation); unit: units on a scale] — The gastrointestinal Symptom Rating Scale (GSRS) is a validated scale, the items range from 1= No discomfort at all to 7= Very severe discomfort.
  The scale ranges from a minimal value of 4 ( No discomfort at all) to a maximum of 28 ( Very severe discomfort)
  units on a scale | 12.6800 (7.11056)
Diarrhea screening [Mean (Standard Deviation); unit: units on a scale] — The gastrointestinal Symptom Rating Scale (GSRS) is a validated scale, the items range from 1= No discomfort at all to 7= Very severe discomfort.
  The scale ranges from a minimal value of 3 ( No discomfort at all) to a maximum of 21 ( Very severe discomfort)
  units on a scale | 10.3200 (5.57315)
Constipation screening [Mean (Standard Deviation); unit: units on a scale] — The gastrointestinal Symptom Rating Scale (GSRS) is a validated scale, the items range from 1= No discomfort at all to 7= Very severe discomfort.
  The scale ranges from a minimal value of 3 ( No discomfort at all) to a maximum of 21 ( Very severe discomfort)
  units on a scale | 7.2000 (4.52769)

OUTCOME MEASURES:

1. Primary Outcome: Gastrointestinal Side Effects and Quality of Life (Total Score of GSRS)
Description: The gastrointestinal Symptom Rating Scale (GSRS) is a validated scale, the items range from 1= No discomfort at all to 7= Very severe discomfort.
  The scale ranges from a minimal value of 15 ( No discomfort at all) to a maximum of 105 ( Very severe discomfort)
  The GSRS contains 15 items, each rated on a seven- point likert scale from no discomfort to very severe discomfort. Based on a factor analysis, the 15 GSRS items breakdown into the following five scales: abdominal ( Abdominal pain, hunger pains and nausea): reflux syndrome (heartburn and acid regurgitation), diarrhea syndrome (diarrhea, loose stools and urgent need for defecation), indigestion syndrome ( borborygmus, abdominal distention, eructation and increased flatus) and constipation syndrome (constipation, hard stools and feeling of incomplete evacuation)
Time Frame: screening, 2, 6 and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liver Transplant Subjects
Number analyzed (Participants) | 29
units on a scale
  screening | 46.000 (21.17585)
  2 weeks | 29.0400 (9.44934)
  6 weeks | 26.2800 (8.79640)
  12 weeks | 25.3600 (8.87356)

2. Primary Outcome: Number of Participants With Cytomegalovirus Infection or Disease
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Liver Transplant Subjects
Number analyzed (Participants) | 29
participants | 0

3. Primary Outcome: Gastrointestinal Side Effects and Quality of Life (-Subscales of GSRS)
Description: The GSRS contains 15 items, each rated on a seven- point likert scale from no discomfort to very severe discomfort. Based on a factor analysis, the 15 GSRS items breakdown into the following five scales: abdominal ( Abdominal pain, hunger pains and nausea): reflux syndrome (heartburn and acid regurgitation), diarrhea syndrome (diarrhea, loose stools and urgent need for defecation), indigestion syndrome ( borborygmus, abdominal distention, eructation and increased flatus) and constipation syndrome (constipation, hard stools and feeling of incomplete evacuation) The range of the scale for abdominal pain was 3 to 21, reflux 2 to 14, diarrhea 3 to 21, indigestion 4 to 28 and constipation 3 to 21.
  Higher values represent more severe discomfort.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liver Transplant Subjects
Number analyzed (Participants) | 29
units on a scale
  Abdominal Pain | 10.78 (5.09)
  Reflux | 2.64 (1.04)
  Indigestion | 7.08 (3.40)
  Diarrhea | 5.44 (3.70)
  Constipation | 4.56 (1.94)

ADVERSE EVENTS:
Time Frame: 0-12 weeks
Description: The protocol specified adverse events including bone marrow suppression, incidence of CMV infection and incidence of acute cellular rejection.
Arm/Group | Liver Transplant Subjects
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No